CLINICAL TRIAL: NCT03504111
Title: PRINT Trial (Platelet Rich Injections vs. Needle Tenotomy): Evaluation of Ultrasound Guided Procedures for the Treatment of Chronic Tendinosis
Brief Title: PRINT Trial (Platelet Rich Injection vs Needle Tenotomy)
Acronym: PRINT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Marissa S. Vasquez, Physician, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB #11064
Record Dates: First submitted 2017-03-30; First posted 2018-04-20 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Lateral Epicondylitis; Tendinosis; Elbow, Tennis; Elbows Tendonitis
MeSH Terms: conditions — Tennis Elbow; Tendinopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Needle Tenotomy (Active Comparator): 1 group will be assigned to get the standard treatment for chronic tendinopathy, percutaneous needle tenotomy (PNT). It is currently considered a standard treatment option. Ultrasound guided PNT with approximately 25 passes through the tendon and enthesis with approximately an 18 gauge needle with adequate amount of anesthetic (lidocaine) for effective anesthesia. Investigators will keep track of the number of passes through the tendon. Investigators will keep track of the amount and type of anesthetic used
  Interventions: Procedure: Percutaneous Needle Tenotomy
- Platelet Rich Plasma (Active Comparator): 1 group will be assigned to the PRP arm. Investigators will have a trained provider draw the blood, and prepare the PRP according to manufacturer and departmental (KP) protocol. Ultrasound guided injection of this PRP using approximately an 18 gauge needle with a single pass through the tendon into affected area as demonstrated on ultrasound. Adequate amount of anesthetic will be given in a separate syringe with adequate amount of anesthetic (lidocaine) for effective anesthesia. Investigators will keep track of amount and type of anesthetic used. The amount of anesthesia will be the same in both arms of the study
  Interventions: Procedure: PRP

INTERVENTIONS:
Procedure: Percutaneous Needle Tenotomy — A sham phlebotomy sample will be drawn on all study participants. Participants in this treatment group will be given local anesthesia with 1% lidocaine and then blinded to the intervention using a blind fold or shielding. Ultrasound guided needle tenontomy with be performed at the common extensor tendon at the area of tendinosis. There will be approximately 25 passes through the tendon with an 18 gauge needle. Investigators will keep track of the number of passes through the tendon. Investigators will keep track of the amount and type of anesthetic used to provide adequate and effective anesthesia
  Other Names: Needle Fenestration
  Arms: Needle Tenotomy
Procedure: PRP — A sham phlebotomy sample will be drawn on all study participants. Participants in this treatment group will be given local anesthesia with 1% lidocaine and then blinded to the intervention using a blind fold or shielding. Ultrasound guided injection of the PRP will be performed at the common extensor tendon at the area of tendinosis. Investigators will keep track of the amount and type of anesthetic used to provide adequate and effective anesthesia to the local skin
  Other Names: Platelet Rich Plasma
  Arms: Platelet Rich Plasma

SUMMARY:
Chronic tendinopathy is often very difficult to treat and causes many patients who suffer from it to have significant pain and loss of function leading to disability. Ultrasound has been shown to be very effective in aiding in the diagnosis of soft tissue disorders including tendinopathy and can help to rule in or out other potential causes that may be confounders. Numerous methods have been tried to treat tendinopathy including rest, NSAIDs, bracing, physical therapy, extracorporal shock wave therapy, anesthetic injections, steroid injections, prolotherapy, nitro patches, surgery and more recently platelet rich plasma, all of which have had conflicting results in the literature. Platelet rich plasma (PRP) is an autologous blood product that contains a high concentration of platelet-derived growth factors that have the potential to enhance healing. In a study by Mishra et al, common extensor tenindosis showed improved pain symptoms (71% vs 55% at 24 weeks) with tenontomy combined with PRP compared to percutaneous needle tenontomy alone. Current studies show conflicting results as to whether PRP improves chronic tendinopathy when compared to steroid injections, and many do not have any control group or comparison group. Percutaneous needle tenotomy is the use of a large gauge needle (18 gauge), which may be performed under ultrasound guidance, to fenestrate repeatedly the area of tendinopathy within a tendon in order to disrupt tendinopathic tissue and to induce bleeding and clot formation with release of growth factors. To date there are no published studies comparing percutaneous needle tenotomy (PNT) alone vs. PRP without concomitant tenotomy. Current literature suggests that needle tenotomy may be superior but no head to head studies are currently found in the literature. Most of the published literature of non-operative treatment of tendinosis does not yield clearly designed trials with clear selection criteria. Current literature also lacks studies with significant number of patients that meet both clinical and ultrasound criteria thus previous studies lack sufficient power. The PRINT TRIAL: may enhance the understanding of a superior treatment if it exists.

Hypothesis: In active adults with chronic tendinopathy who have failed to respond to standard of care treatment, the use of ultrasound guided percutaneous needle tenotomy (PNT) alone is superior to PRP without concomitant tenotomy.

DETAILED DESCRIPTION:
The objective of our study is to determine if percutaneous needle tenontomy is superior to platelet rich plasma for the treatment of chronic tendinosis. Diagnosis of tendinosis will be confirmed utilizing ultrasound diagnostic criteria similar to past published studies. The study will be a prospective single blinded study utilizing sham phlebotomy, which currently is not found in the published literature. All interventions will be done ultrasound-guided which no studies in the published literature have done prospectively. The main variables of interest include patient outcomes such as improved function, objective clinical improvement as seen on serial ultrasound surveillance and patient reported utility. Secondary outcomes include: determine patient's ability to return to sport or activity and level of activity able to achieve using validated questionnaires. Lastly, compliance with survival curve data will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Adults: 18 years and older
* Diagnosed with: Lateral epicondylitis or common extensor tendinopathy
* Has had symptoms for more than 3 months
* Failed conservative treatment with an eccentric loading protocol that was formally taught and attempted for at least 6 weeks.
* Failed at least 1 corticosteroid injection (anatomically or ultrasound guided injection)

Exclusion Criteria:

* Age less than 18 years
* Pregnant or breast feeding females
* Previous surgery to the area of interest
* Previous needling procedure to the area of interest in the last 3 months
* Previous steroid injection to the area of interest in the last 3 months
* Previous PRP or autologous blood or prolotherapy to the area of interest
* Patients treated for a Workers Compensation related injury
* Any systemic disease that may play a causative role or delay in healing such as rheumatoid arthritis, lupus, immunodeficiency
* Severe degenerative bone disease or severe vascular disease that may be a confounder

Diagnosis of concomitant nerve involvement in area of interest:

* Carpal tunnel, radial nerve impingement, cervical radiculopathy in patients with lateral epicondylitis
* Any contraindication to use of lidocaine or injections
* Will record if patient is taking any medications that may alter bleeding or clotting such as aspirin, Plavix, Coumadin, Aggrenox, heparin, lovenox, etc, but this will be a relative contraindication and decision is made by patient and provider after informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in DASH Symptoms Score | Change in symptom score between pre-study and 1 year
  Disabilities of the arms, shoulder and hand symptoms questionnaire and score

CONTACTS AND LOCATIONS:
Overall Officials: Marissa S Vasquez, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- KP-LAMC, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abate M, Verna S, Di Gregorio P, Salini V, Schiavone C. Sonographic findings during and after Platelet Rich Plasma injections in tendons. Muscles Ligaments Tendons J. 2014 May 8;4(1):29-34. eCollection 2014 Jan. PMID 24932444
- [Background] Finnoff JT, Fowler SP, Lai JK, Santrach PJ, Willis EA, Sayeed YA, Smith J. Treatment of chronic tendinopathy with ultrasound-guided needle tenotomy and platelet-rich plasma injection. PM R. 2011 Oct;3(10):900-11. doi: 10.1016/j.pmrj.2011.05.015. Epub 2011 Aug 26. PMID 21872551
- [Background] Mishra A, Pavelko T. Treatment of chronic elbow tendinosis with buffered platelet-rich plasma. Am J Sports Med. 2006 Nov;34(11):1774-8. doi: 10.1177/0363546506288850. Epub 2006 May 30. PMID 16735582
- [Background] Chiavaras MM, Jacobson JA. Ultrasound-guided tendon fenestration. Semin Musculoskelet Radiol. 2013 Feb;17(1):85-90. doi: 10.1055/s-0033-1333942. Epub 2013 Mar 13. PMID 23487340
- [Background] Hamilton BH, Best TM. Platelet-enriched plasma and muscle strain injuries: challenges imposed by the burden of proof. Clin J Sport Med. 2011 Jan;21(1):31-6. doi: 10.1097/JSM.0b013e318205a658. PMID 21200168
- [Background] Boyer MI, Hastings H 2nd. Lateral tennis elbow: "Is there any science out there?". J Shoulder Elbow Surg. 1999 Sep-Oct;8(5):481-91. doi: 10.1016/s1058-2746(99)90081-2. PMID 10543604
- [Background] Paoloni J, De Vos RJ, Hamilton B, Murrell GA, Orchard J. Platelet-rich plasma treatment for ligament and tendon injuries. Clin J Sport Med. 2011 Jan;21(1):37-45. doi: 10.1097/JSM.0b013e31820758c7. PMID 21200169
- [Background] Balasubramaniam U, Dissanayake R, Annabell L. Efficacy of platelet-rich plasma injections in pain associated with chronic tendinopathy: A systematic review. Phys Sportsmed. 2015 Jul;43(3):253-61. doi: 10.1080/00913847.2015.1005544. Epub 2015 Jan 20. PMID 25599747
- [Background] Foster TE, Puskas BL, Mandelbaum BR, Gerhardt MB, Rodeo SA. Platelet-rich plasma: from basic science to clinical applications. Am J Sports Med. 2009 Nov;37(11):2259-72. doi: 10.1177/0363546509349921. PMID 19875361
- [Background] Housner JA, Jacobson JA, Misko R. Sonographically guided percutaneous needle tenotomy for the treatment of chronic tendinosis. J Ultrasound Med. 2009 Sep;28(9):1187-92. doi: 10.7863/jum.2009.28.9.1187. PMID 19710216
- [Background] McShane JM, Shah VN, Nazarian LN. Sonographically guided percutaneous needle tenotomy for treatment of common extensor tendinosis in the elbow: is a corticosteroid necessary? J Ultrasound Med. 2008 Aug;27(8):1137-44. doi: 10.7863/jum.2008.27.8.1137. PMID 18645071
- [Background] Mautner K, Colberg RE, Malanga G, Borg-Stein JP, Harmon KG, Dharamsi AS, Chu S, Homer P. Outcomes after ultrasound-guided platelet-rich plasma injections for chronic tendinopathy: a multicenter, retrospective review. PM R. 2013 Mar;5(3):169-75. doi: 10.1016/j.pmrj.2012.12.010. Epub 2013 Feb 9. PMID 23399297
- [Background] Mautner K, Kneer L. Treatment of tendinopathies with platelet-rich plasma. Phys Med Rehabil Clin N Am. 2014 Nov;25(4):865-80. doi: 10.1016/j.pmr.2014.06.008. Epub 2014 Aug 30. PMID 25442163
- [Background] Sanchez M, Anitua E, Orive G, Mujika I, Andia I. Platelet-rich therapies in the treatment of orthopaedic sport injuries. Sports Med. 2009;39(5):345-54. doi: 10.2165/00007256-200939050-00002. PMID 19402740
- [Background] Sims SE, Miller K, Elfar JC, Hammert WC. Non-surgical treatment of lateral epicondylitis: a systematic review of randomized controlled trials. Hand (N Y). 2014 Dec;9(4):419-46. doi: 10.1007/s11552-014-9642-x. PMID 25414603
- [Derived] Karjalainen TV, Silagy M, O'Bryan E, Johnston RV, Cyril S, Buchbinder R. Autologous blood and platelet-rich plasma injection therapy for lateral elbow pain. Cochrane Database Syst Rev. 2021 Sep 30;9(9):CD010951. doi: 10.1002/14651858.CD010951.pub2. PMID 34590307